CLINICAL TRIAL: NCT03517878
Title: A Non-randomized Comparative Cohort Study Evaluating a Home-based Community Health Worker Program in the Rural Eastern Cape Province of South Africa
Brief Title: Evaluation of a Home-based Community Health Worker Program in Rural Eastern Cape, South Africa
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Collaborators: The ELMA Foundation (Other); University of Stellenbosch (Other); Philani Maternal Child Health and Nutrition Project (Unknown)
Responsible Party: Sponsor
Other Study IDs: N14/03/019
Record Dates: First submitted 2018-03-14; First posted 2018-05-08 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2018-10

CONDITIONS: HIV Infections; HIV/AIDS; Depression; Depressive Symptoms; Alcohol Use Disorder; Alcohol Drinking; Stunting; Alcohol; Harmful Use; Child Development; Child Malnutrition; Child Nutrition Disorders; Birth Weight Less Than 10Th Percentile
Keywords: Community Health Worker; Pregnancy; Breast Feeding; Child Development; Home Visits; Infants
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; Depression; Alcoholism; Alcohol Drinking; Growth Disorders; Child Nutrition Disorders; Breast Feeding

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Comprehensive CHW Cohort: Pregnant women who become mothers and their infants living in areas served by the comprehensive CHW program. These are areas around two primary health care clinics and matched to the Control Cohort clinic areas.
  Interventions: Behavioral: Comprehensive CHW Program
- Control Cohort: Pregnant women who become mothers and their infants living in areas that are not served by the comprehensive CHW program. These are areas around two primary health care clinics and matched to the Comprehensive CHW Cohort clinic areas.

INTERVENTIONS:
Behavioral: Comprehensive CHW Program — The comprehensive CHW Cohort will receive home visits from CHWs recruited, trained, and supervised by the Philani organization. Philani has a 30-year history of non-stigmatizing home-based support for women and children in Cape Town. The organization has been operating their comprehensive CHW program in the rural Eastern Cape since 2010; however, in the research areas, CHWs have only been active for one year prior to initiation of the study. Philani recruits CHWs that are "positive peer deviants" to serve as role models in the community. The CHWs then receive training, materials, and skills to address major community health challenges of HIV, TB, malnutrition, alcohol use, and depression. The CHWs also receive ongoing monitoring and supervision as well as support for difficult cases.
  Groups: Comprehensive CHW Cohort

SUMMARY:
The purpose of this early Phase 2 comparison trial is to evaluate the impact of community health worker (CHW) home visitors on pregnant women and their children in a rural setting in the rural Eastern Cape of South Africa. The intervention provided by the CHWs targets underweight children, mothers living with HIV (MLH), mothers using alcohol, and depressed mothers with the goal of supporting pregnant women to improve birth outcomes, decrease the number of children born with a low birthweight, and develop child caretaking skills over time. UCLA has identified and matched four areas surrounding primary health care clinics: two intervention areas in which this CHW program has been running for one year, and two control areas without the program. Mothers in the research area are followed for one year after giving birth.

DETAILED DESCRIPTION:
Inequalities in the quality and accessibility of healthcare between urban centers and rural areas is a global challenge that is particularly stark for low and middle-income countries (LMIC). Maternal and child health (MCH) in rural South Africa is negatively impacted by large distances, poor infrastructure, and a shortage of healthcare workers at clinics and hospitals.

Home visiting has been repeatedly demonstrated efficacious in addressing some of these challenges and improving MCH outcomes, including when delivered by CHW in LMIC. However, there is limited research on the effectiveness of implementing these types of programs in rural areas.

The investigators have shown that with training, supervision, and accountability, CHW home visits are effective in improving MCH over the first five years of life. These results were observed in a successful randomized controlled trial conducted in peri-urban townships in Cape Town, South Africa. CHW were trained to address HIV, alcohol, and malnutrition among all pregnant women in a neighborhood, to avoid stigma, and to address multiple health challenges concurrently. The visits significantly improved MCH outcomes over five years. Based on these results, this comprehensive CHW home visiting program served as one model for re-engineering primary health care to include 65,000 paraprofessionals providing home-based care in South Africa.

This early phase two comparison trial examines whether the same comprehensive CHW home visiting program can be effectively implemented in a deeply rural area of the Eastern Cape in South Africa. Two matched cohorts of women and their children, one in areas where the comprehensive CHW program has been active for one year and one in areas without the program, will be followed from pregnancy through the first 12 months after giving birth. Stellenbosch University interviewers will independently assess outcomes of each mother at pregnancy, and of the mothers and infants within two weeks of post-birth, 6 months, and 12 months later. The primary outcomes are a combined measures of maternal and child health including maternal HIV testing, depression, and alcohol use, as well as the child's nutrition, physical growth, development, and healthcare and a measure of how MLH comply with tasks for PMTCT.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who are or become mothers living in the catchment area at the time of recruitment
* Women not identified as psychotic or delusional based on the interviewer's judgment
* Women able to provide informed consent

Exclusion Criteria:

* Inability to give informed consent
* Inability to converse with the interviewer or the CHW
* Miscarriage or stillbirth
* Death of the infant
* Death of the mother

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Cohorts include all women meeting inclusion criteria from the catchment areas surrounding four clinics in the rural Eastern Cape.
Sampling Method: Non-Probability Sample
Enrollment: 1490 (Actual)
Dates: Start 2014-08-11 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Composite outcome: Number of significantly improved child and maternal outcomes | 12 months
  Out of 11 variables, we run 1000 simulations on the distribution of 0 and 1. The investigators total number of outcomes (each scored as 0=not present or 1=present) and determine if the Comprehensive CHW Cohort sum is significantly greater than expected based on the Control Cohort.
  For Mothers:
  1. Breastfeeding
  2. No alcohol in pregnancy
  3. Not depressed
  4. Adhere to medical regimens
     * For all mothers:
       -4 antenatal care visits
     * For HIV+ mothers:
       * Test for HIV
       * Take ARV
       * Give infant NVP and bactrim
       * infant PCR
       * exclusive breastfeeding
     For Children:
  5. Not low birth weight
  6. Growth in height
  7. Growth in weight
  8. Hospitalizations
  9. Developmental milestones
  10. Vaccinations
  11. Child support grant
  Harwood JM, Weiss RE, Comulada WS. Beyond the Primary Endpoint Paradigm: A Test of Intervention Effect in HIV Behavioral Intervention Trials with Numerous Correlated Outcomes. Prevention Science. 2017 Jul 1;18(5):526-33.

SECONDARY OUTCOMES:
Breastfeed for three months | 6 months, 12 months
  Mothers are asked at the 6 month and 12 month follow up "How long after your baby's birth did you stop breastfeeding your baby completely?"
Breastfeed for six months | 6 months, 12 months
  Mothers are asked at the 6 month and 12 month follow up "How long after your baby's birth did you stop breastfeeding your baby completely?"
No alcohol after learning that the participant was pregnant | Birth
  At the birth interview mothers are asked "Have you ever used alcohol during this pregnancy?" and follows up with "Did you continue to drink alcohol after you knew you were pregnant?"
Attend 4 antenatal care visits | Birth
  At the birth interview antenatal care cards are inspected and mothers are asked "How many antenatal care visits did you attend?"
Not depressed, EPDS below 13 | Birth, 6 months, 12 months
  EPDS is asked after birth, 6 months after birth, and at 12 months after birth.
Infant was not low birth weight | Birth
  Birth weight is recorded from child's road to health card and baby is weighed by data collector shortly after birth (this value is used when road to health card is not available).
Growth in height-for-age (above -2SD) | Birth, 6 months, 12 months
  Child height/length is recorded shortly after birth, at 6 months, and at 12 months. Values are compared to WHO norms and turned into a Z score.
Growth in weight-for-age (above -2SD) | Birth, 6 months, 12 months
  Child weight is recorded shortly after birth, at 6 months, and at 12 months. Values are compared to WHO norms and turned into a Z score.
Number of Hospitalizations | 6 months, 12 months
  At 6 months and 12 months after birth mothers are asked "During the past 3 months, have you taken the child to the hospital for any reason?" and "How many times have you taken the child to the hospital?"
WHO developmental scale measures at 50th percentile | 12 months
  WHO measures of child development are used and children are compared to the mean level of achievement for their age. Fussy or sleepy children may be unable to be evaluated.
Vaccinations up to date | 12 months
  Data collectors examine the child's road to health card to determine if all immunizations are up to date and which ones are missing. A photo is taken of this page for confirmation.
Has Child Support Grant | 12 months
  Mothers are asked "Does the child get a child support grant?"
Mothers test for HIV during pregnancy | Birth
  Data collectors look for any evidence on the antenatal card of an HIV test during pregnancy. If not, or if card is unavailable, check with the mother if she has previously tested positive for HIV or ask "Did you have a test for HIV during this pregnancy?"
MLH take ARV during pregnancy | 12 months
  Mothers are asked "When did you start taking ARVs?" and antenatal cards and health cards are examined for evidence of ARV prescription and start date.
Give infant NVP and Bactrim | 6 months
  Mothers are asked "Did you get Nevarapine syrup for your baby around the time of birth?"; "Are you currently using nevirapine syrup for the baby?" and "Are you currently still giving your child bactrim?"
PCR testing at 6 weeks | 12 months
  Mothers are asked "Has you child been tested for HIV yet?" and "Do you know what the result of your child's HIV test (PCR) is?" Data collectors independently confirm this information on the child's road to health card to determine how many times (if at all) the child has been tested for HIV?
6 months exclusive breastfeeding | 6 months
  Mothers are asked "How soon after birth did you give your child something else in addition to breastmilk?" In addition, mothers are asked to provide a 24 hour, 1 months, and 3 month dietary recall.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Tomlinson, PhD, Principal Investigator — University of Stellenbosch; Karl W le Roux, MB ChB, Principal Investigator — Zithulele Hospital; Ingrid le Roux, MD, Principal Investigator — Philani Maternal Child Health and Nutrition Project
Locations (2):
- South Africa (2):
  - Zithulele Hospital, Mqanduli, Eastern Cape
  - Stellenbosch University, Stellenbosch

REFERENCES:
- See also: Philani Website — http://www.philani.org.za/